CLINICAL TRIAL: NCT06006507
Title: The Effect of Exercise on Menstrual Symptoms: a Randomised Controlled Trial
Brief Title: The Effect of Exercise on Menstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar58
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Menstrual Problem
Keywords: sleep; menstruation; stress
MeSH Terms: conditions — Menstruation Disturbances | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise treatments
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): no exercise will be given
  Interventions: Other: control
- exercise group (Experimental): exercise training will be given and they will be asked to exercise regularly.
  Interventions: Other: exercise

INTERVENTIONS:
Other: control — no exercise will be given
  Arms: control group
Other: exercise — In line with the recommendation of the World Health Organization, the exercise group will do 150 minutes of moderate-intensity walking a week and strengthening exercises prepared by the physiotherapist two days a week. Strengthening exercises will be taught by the physiotherapist in a session with the people in the exercise group in groups of five, and then exercise lists will be given to the people on digital exercise platform, where there are video narrations of the exercises. In addition, the participants will be asked to do balance exercises and macular exercise.
  Arms: exercise group

SUMMARY:
The aim of this study is to contribute to the determination of the relationship between exercise and menstrual symptoms and to create an alternative for non-pharmacological coping methods with menstrual symptoms.

DETAILED DESCRIPTION:
The type of research is randomized controlled trial. An average of 50 people who do not have exercise habits will participate in the study, and two randomized groups will be formed as exercise group and control group. Everyone will be asked to fill in the Menstruation Symptom Scale, the Menstruation Distress Scale, the Pittsburgh Sleep Quality Scale, the Fatigue Severity Scale, the International Physical Activity Scale, the Personal Information Form prepared by us, and the Voluntary and Consent Form during their menstrual period. The duration of the study will cover 3 (three) menstrual periods of the individuals. At the beginning and end of the study; They will be asked to fill in the Pittsburgh Sleep Quality Scale, Fatigue severity scale, International Physical Activity Questionnaire Short form, Menstruation Symptom Scale and Menstruation Distress Complaint List.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-50 whose menstrual cycle continues,
* Those who have emotional or physical problems during menstruation periods,
* Those whose menstrual cycle is between 21-40 days on average

Exclusion Criteria:

* Those with chronic disease
* Those with a diagnosed gynecological disease,
* Those who receive any medical treatment,
* Persons with dysmenorrhea and anemia.
* People who exercise regularly.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — menstrual cycle Female only
Enrollment: 54 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Scale | 14 weeks
  The pittsburgh Sleep Quality Index is a quantitative measure of sleep quality to define good and bad sleep. It includes 24 questions in total. The self-assessment questions include various items related to sleep quality. The total score is between 0-21. A high total score indicates poor sleep quality. The index does not indicate the presence of sleep disturbances or the prevalence of sleep disturbances. However, a pittsburgh Sleep Quality Index total score of five or more indicates poor sleep quality.
Fatigue Severity Scale | 14 weeks
  It consists of 9 questions. Each question is scored between 1 and 7. Statements Regarding Scoring 1. I strongly disagree 3. I tend to disagree 5. I tend to agree 2. I disagree 4. I am undecided 6. I agree 7. I strongly agree. ) the score of the answers given to the question is added and divided by 9. If the result is less than 2.8, it is evaluated as "no fatigue". If the result is greater than 6.1, it is considered as "chronic fatigue syndrome".
Short form of the International Physical Activity Questionnaire | 14 weeks
  provides information on time spent walking, moderate and vigorous activities, and time spent sitting. Calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. The energy required for activities is calculated with the metabolic equivalent(MET) -minute score. Standard metabolic equivalent (MET) values have been established for these activities.
Menstruation Symptom Scale | 14 weeks
  It is a 5-point Likert-type scale and consists of three sub-parameters: 'negative effects/somatic effects', 'menstrual pain' and 'coping methods', and 22 items. The person is asked to give a score between '1' never and '5' always for the symptoms they experience related to menstruation. The Menstruation Symptom Scale (MSS) score is calculated by taking the total score average. An increase in the mean score indicates an increase in the severity of menstrual symptoms.
Menstruation Distress Complaints List | 14 weeks
  He questions the severity of these symptoms one week before the menstruation, during the last menstruation, and on other days. Complaints are scored from 0 to 4. These are 0: no symptoms, 1: little, 2: moderate, 3: severe, and 4: very severe. The lowest score that can be obtained from the scale is 0 for each term, and the highest score is 188.

CONTACTS AND LOCATIONS:
Overall Officials: Merve KOÇAK, Study Chair — Bahçeşehir University
Locations (1):
- Üsküdar Unıversıty, Beşiktaş, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eccleston CA, Goldenholz SR, Goldenholz DM. Exercise, medication adherence, and the menstrual cycle: How much do these change seizure risk? Epilepsy Res. 2022 Dec;188:107052. doi: 10.1016/j.eplepsyres.2022.107052. Epub 2022 Nov 15. PMID 36403515
- [Result] Janse de Jonge XA. Effects of the menstrual cycle on exercise performance. Sports Med. 2003;33(11):833-51. doi: 10.2165/00007256-200333110-00004. PMID 12959622
- [Result] Oosthuyse T, Bosch AN. The effect of the menstrual cycle on exercise metabolism: implications for exercise performance in eumenorrhoeic women. Sports Med. 2010 Mar 1;40(3):207-27. doi: 10.2165/11317090-000000000-00000. PMID 20199120
- [Result] Pereira HM, Larson RD, Bemben DA. Menstrual Cycle Effects on Exercise-Induced Fatigability. Front Physiol. 2020 Jun 26;11:517. doi: 10.3389/fphys.2020.00517. eCollection 2020. PMID 32670076
- [Result] Nie J, Zhang H, Kong Z, Wang C, Liu Y, Shi Q, George K. The impact of exercise modality and menstrual cycle phase on circulating cardiac troponin T. J Sci Med Sport. 2020 Mar;23(3):309-314. doi: 10.1016/j.jsams.2019.10.003. Epub 2019 Oct 10. PMID 31690491
- [Derived] Kocak M, Sevgin O. The effect of exercise on menstrual symptoms: a randomized controlled trial. BMC Womens Health. 2025 Aug 23;25(1):406. doi: 10.1186/s12905-025-03940-8. PMID 40849627